CLINICAL TRIAL: NCT06554496
Title: Obstructive Sleep Apnea Severity and Xanthine Oxidoreductase Activity: Mechanisms and Clinical Implications
Brief Title: XOR Levels in OSA Patients (XOR-OSA)
Acronym: XOR-OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Principal Investigator, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-629
Record Dates: First submitted 2024-08-06; First posted 2024-08-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Xanthine Oxidoreductase; CPAP treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP Treatment Group (Experimental): Patients with Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) who are eligible for Continuous Positive Airway Pressure (CPAP) therapy.
  Interventions: Device: CPAP Treatment

INTERVENTIONS:
Device: CPAP Treatment — Continuous Positive Airway Pressure (CPAP) therapy will be administered to patients for 3 months. The CPAP device will be set to deliver a continuous flow of air at a prescribed pressure to keep the patient's airway open during sleep.

SUMMARY:
The level of xanthine oxidoreductase (XOR) in plasma is associated with oxidative stress and inflammation. Obstructive Sleep Apnea (OSA) is characterized by repeated upper airway obstruction and apneas during sleep, leading to chronic intermittent hypoxemia. The specific role of XOR in OSA, its relationship with the severity of OSA, and the changes in XOR levels before and after CPAP treatment remain unclear. The study will enroll 80 patients from the First Affiliated Hospital of Nanjing Medical University, categorized by their Apnea-Hypopnea Index (AHI) into mild, moderate, and severe OSA groups. Participants will undergo baseline assessments including polysomnography (PSG) and measurements of XOR activity and biomarkers such as uric acid, endothelin-1 (ET-1), endothelial nitric oxide synthase (eNOS), and inflammatory markers. Eligible patients will receive CPAP treatment for 3 months, after which their XOR activity and biomarker levels will be re-evaluated to assess treatment efficacy.

DETAILED DESCRIPTION:
Xanthine oxidoreductase (XOR) is an enzyme involved in the oxidative metabolism of purines, producing reactive oxygen species (ROS) as byproducts. Elevated XOR activity is associated with increased oxidative stress and inflammation. In patients with Obstructive Sleep Apnea(OSA), repeated episodes of hypoxia and reoxygenation lead to oxidative stress and inflammatory responses. However, the specific changes in XOR activity in OSA patients are not well understood.

This study aims to evaluate the effects of Continuous Positive Airway Pressure (CPAP) treatment on patients with OSA by analyzing XOR activity and related biomarkers. The primary objective is to assess the correlation between XOR activity levels and the severity of OSA, and to determine how these levels change following a 3-month CPAP intervention.

The study will enroll 80 patients aged 18-80 years from the First Affiliated Hospital of Nanjing Medical University. Participants will be diagnosed with OSA according to established guidelines, and must be first-time visitors with no prior OSA surgery or CPAP treatment history. Patients with severe cerebrovascular diseases, psychiatric conditions, diagnosed diabetes with significant vascular complications, severe COPD, pulmonary hypertension, heart failure, or pregnancy will be excluded.

All participants will undergo polysomnography (PSG) to determine the Apnea-Hypopnea Index (AHI) and categorize them into mild, moderate, or severe OSA groups.

Blood samples will be collected to measure baseline XOR activity and related biomarkers, including uric acid, endothelin-1 (ET-1), endothelial nitric oxide synthase (eNOS), C-reactive protein (CRP), tumor necrosis factor-alpha (TNF-α), interleukin-6 (IL-6), malondialdehyde (MDA), superoxide dismutase (SOD), hypoxia-inducible factor-1 (HIF-1), and angiotensin II (Ang II).

Eligible patients will receive CPAP therapy for a duration of 3 months. Patients unsuitable for CPAP therapy will receive alternative treatments such as upper airway surgery, oral appliances, or weight reduction programs. After 3 months of CPAP therapy, participants will undergo follow-up PSG to reassess sleep parameters. Blood samples will be collected again to measure changes in XOR activity and related biomarkers.

The data collected will be analyzed using SPSS software. Correlation analysis will be performed to assess the relationship between AHI, lowest SpO2, oxygen load, blood pressure load, ESS sleepiness scores, and XOR levels. Paired t-tests will be used to compare pre- and post-treatment XOR activity and biomarker levels. Repeated measures ANOVA will be conducted to evaluate the long-term changes and sustained effects of CPAP therapy.

This study aims to provide a comprehensive understanding of the biochemical impacts of CPAP therapy on patients with OSAHS. The findings are expected to identify potential biomarkers for assessing treatment efficacy and to guide future therapeutic strategies, ultimately improving patient outcomes in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 80 years.
2. Diagnosed with Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS)(apnea-hypopnea index≥5/h).
3. First-time diagnosis, with no previous surgical interventions or CPAP treatment for OSA.
4. Ability and willingness to provide informed consent for participation in the study.

Exclusion Criteria:

1. History of severe stroke or cerebral hemorrhage, or presence of neurological or psychiatric conditions that could affect study results.
2. Presence of active malignancies or other severe underlying diseases, such as severe liver or kidney dysfunction. Diagnosed with diabetes or other significant vascular diseases.
3. Presence of severe chronic obstructive pulmonary disease (COPD), severe asthma, severe pulmonary hypertension, or heart failure caused by any condition.
4. Pregnancy or having other conditions that make participation in this study unsuitable.
5. Extremely debilitated patients or those with severe underlying conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Xanthine Oxidoreductase (XOR) Activity | Baseline and 3 months of CPAP therapy
  To measure changes in XOR activity levels in OSA patients with different severities, using enzyme-linked immunosorbent assay (ELISA) techniques, before and after 3 months of CPAP therapy, reported in units per liter (U/L).
Apnea-Hypopnea Index (AHI) | Baseline and 3 months of CPAP therapy.
  To measure changes in the Apnea-Hypopnea Index, quantifying the severity of sleep apnea, reported as the number of apneas and hypopneas per hour of sleep.

SECONDARY OUTCOMES:
Uric Acid Levels | Baseline and 3 months of CPAP therapy
  Assess changes in serum uric acid levels, reported in milligrams per deciliter (mg/dL), using ELISA.
Endothelial Nitric Oxide Synthase (eNOS) Activity | Baseline and 3 months of CPAP therapy
  Measure changes in eNOS activity in serum, reported in units per liter (U/L), using ELISA.
C-Reactive Protein (CRP) Levels | Baseline and 3 months of CPAP therapy
  Measure changes in C-reactive protein levels in serum, reported in milligrams per liter (mg/L), using ELISA.
Superoxide Dismutase (SOD) Activity | Baseline and 3 months of CPAP therapy.
  Assess changes in superoxide dismutase activity in serum, reported in units per milliliter (U/mL), using ELISA.
Time with Oxygen Saturation Below 90% (T90%) | Baseline and 3 months of CPAP therapy.
  To measure the duration of time spent with oxygen saturation levels below 90% during sleep, reported as a percentage of total sleep time with SpO2 below 90%.
Subjective Sleepiness | Baseline and 3 months of CPAP therapy.
  To assess changes in subjective sleepiness using the Epworth Sleepiness Scale (ESS), which is a self-administered questionnaire. The ESS measures the general level of daytime sleepiness, or average sleep propensity in daily activities, on a scale ranging from 0 to 24. A higher score on this scale indicates a greater likelihood of falling asleep in a variety of situations, suggesting worse daytime sleepiness.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared. The informed consent will be ansigned before enrolled in the study and ensured to keep personal information confidential.

REFERENCES:
- [Result] Bortolotti M, Polito L, Battelli MG, Bolognesi A. Xanthine oxidoreductase: One enzyme for multiple physiological tasks. Redox Biol. 2021 May;41:101882. doi: 10.1016/j.redox.2021.101882. Epub 2021 Jan 27. PMID 33578127
- [Result] Saugstad OD. Role of xanthine oxidase and its inhibitor in hypoxia: reoxygenation injury. Pediatrics. 1996 Jul;98(1):103-7. PMID 8668378
- [Result] Ali MH, Schlidt SA, Chandel NS, Hynes KL, Schumacker PT, Gewertz BL. Endothelial permeability and IL-6 production during hypoxia: role of ROS in signal transduction. Am J Physiol. 1999 Nov;277(5):L1057-65. doi: 10.1152/ajplung.1999.277.5.L1057. PMID 10564193
- [Result] Vickneson K, George J. Xanthine Oxidoreductase Inhibitors. Handb Exp Pharmacol. 2021;264:205-228. doi: 10.1007/164_2020_383. PMID 32789757
- [Result] Nguyen NH, Tran GB, Nguyen CT. Anti-oxidative effects of superoxide dismutase 3 on inflammatory diseases. J Mol Med (Berl). 2020 Jan;98(1):59-69. doi: 10.1007/s00109-019-01845-2. Epub 2019 Nov 13. PMID 31724066